CLINICAL TRIAL: NCT04863885
Title: Phase I/II Study of Ipilimumab Plus Nivolumab (IPI-NIVO) Combined With Sacituzumab Govitecan (SG)as First-line Treatment for Cisplatin-ineligible Metastatic Urothelial Carcinoma
Brief Title: Combination of Ipi/Nivo Plus Sacituzumab Govitecan in Metastatic Cisplatin Ineligible Urothelial Carcinoma Patients
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry); Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MCC-20943; CA209-63Y (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2021-04-26; First posted 2021-04-28 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Urothelial Carcinoma
Keywords: mUC; Bladder cancer
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms | interventions — Ipilimumab; Nivolumab; sacituzumab govitecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1 Dose Level 1 (Experimental): Participants will be treated at dose level 1: Ipilumumab 3mg/kg + Nivolumab 1mg/kg IV day 1 every 3 weeks for 4 cycles, followed by Nivolumab 360 mg every 3 weeks. Sacituzumab Govitecan 8 mg/kg IV will be administered days 1 and 8 every 3 weeks.
  Interventions: Drug: Ipilimumab; Drug: Nivolumab; Drug: Sacituzumab govitecan
- Phase 1 Dose Level 2 (Experimental): Participants will be treated at dose level 2: Ipilumumab 3mg/kg + Nivolumab 1mg/kg IV day 1 every 3 weeks for 4 cycles, followed by Nivolumab 360 mg every 3 weeks. Sacituzumab Govitecan 10 mg/kg IV will be administered days 1 and 8 every 3 weeks.
  Interventions: Drug: Ipilimumab; Drug: Nivolumab; Drug: Sacituzumab govitecan
- Phase 1 Dose Level -1 (Experimental): If dose reduction is indicated, participants will be treated at dose level -1: Ipilumumab 3mg/kg + Nivolumab 1mg/kg IV day 1 every 3 weeks for 4 cycles, followed by Nivolumab 360 mg every 3 weeks. Sacituzumab Govitecan 6 mg/kg IV will be administered days 1 and 8 every 3 weeks
  Interventions: Drug: Ipilimumab; Drug: Nivolumab; Drug: Sacituzumab govitecan
- Phase 2: Treatment at Maximum Tolerated Dose (MTD) (Experimental): Participants will be treated at with Ipilumumab 3mg/kg + Nivolumab 1mg/kg IV day 1 every 3 weeks for 4 cycles, followed by Nivolumab 360 mg every 3 weeks plus the maximum tolerated dose of Sacituzumab Govitecan days 1 and 8 every 3 weeks.
  Interventions: Drug: Ipilimumab; Drug: Nivolumab; Drug: Sacituzumab govitecan

INTERVENTIONS:
Drug: Ipilimumab — Participants will receive Ipilimumab 3 mg/kg
  Other Names: Yervoy
Drug: Nivolumab — Participants will receive Nivoumab 1mg/kg
  Other Names: Opdivo
Drug: Sacituzumab govitecan — Participants will be treated at 1 of 2 dose levels of Sacituzumab govitecan, either at 8 mg/kg, 10 mg/kg, or 6 mg/kg.
  Other Names: Trodelvy

SUMMARY:
The purpose of this study is to see how well the study drugs called Ipilimumab plus Nivolumab (IPI-NIVO) work when added to another study drug called Sacituzumab Govitecan for people who have metastatic bladder cancer.

DETAILED DESCRIPTION:
The phase I component of this study will evaluate fixed doses of ipilimumab and nivolumab (3 mg/kg and 1 mg/kg, respectively) IV every 3 weeks x 4 cycles combined with a starting dose of sacituzumab govitecan Level 1 of 8 mg/kg IV days 1,8 every 3 weeks (1 cycle) x 4 cycles. One dose escalation to 10 mg/kg and one dose reduction to dose level minus 1 of sacituzumab govitecan 6 mg/kg days 1,8 every 3 weeks is allowed.

The phase II component will be conducted as two-stage trial enrolling 34 patients with a futility interim analysis after stage 1 (13 patients). After 4 cycles, patients will continue maintenance nivolumab 360 mg IV every Q 21 days along with RP2 dose of SG D1,8 Q21 days till progression of disease or intolerable toxicities or patient decision. Radiographic imaging is performed every 12 weeks to assess response.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Able to understand and give written informed consent.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Participants with histologically documented locally advanced or metastatic urothelial carcinoma. Upper and lower tract tumors are permitted and mixed histologies are permitted if urothelial carcinoma is the predominant histology (≥50%).
* Ineligiblity for cisplatin-based chemotherapy, defined by any of the following: (a) Creatinine clearance (CL) <60 mL/min. GFR should be calculated from serum/plasma creatinine using the Cockcroft-Gault formula. (b) CTCAE v5.0 Grade > 1 hearing loss (c) CTCAE v5.0 Grade > 1 neuropathy (d) NYHA Class > II cardiac dysfunction
* Adequate organ function laboratory values as defined per protocol
* Have measurable disease by CT or MRI as per RECIST 1.1 criteria. Tumor lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre- menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply: (a) Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy). (b) Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
* Male participants must agree to use an adequate method of contraception starting with the first dose of study therapy through 7 months after the last dose of study therapy. Female participants if sexually active must agree to use dual methods of contraception during the study and for a minimum period of 5 months after the last dose of study drug.

Exclusion Criteria:

* Women who are pregnant or lactating.
* Currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks prior to the first dose of trial treatment.
* Prior chemotherapy for metastatic urothelial carcinoma at any time in the patient's medical history.
* Small-cell carcinoma component
* Prior chemotherapy for localized urothelial carcinoma completed within 12 months before registration. Has received anti-PD-1/PD-L1 therapy previously, except if used in earlier stage urothelial carcinoma such as non-muscle invasive bladder cancer (NMIBC) or muscle invasive bladder cancer (MIBC) as neoadjuvant or adjuvant therapy and completed >3 months prior to registration.
* Prior therapy with sacituzumab govitecan, irinotecan, or any topoisomerase I-containing regimen or antibody-drug conjugate
* Received radiation therapy for bone metastasis ≤2 weeks, any other radiation therapy within 4 weeks before first dose of study treatment. Systemic treatment with radionuclides within 6 weeks before the first dose of study treatment. Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Requires concomitant medication interfering with ABCA1 transporter or UGT1A1
* Participants with Gilbert's disease.
* An active second malignancy. Note: Participants with a history of malignancy that has been completely treated, with no evidence of active cancer for 3 years prior to enrollment, or subjects with surgically cured tumors with low risk of recurrence are allowed to- enroll.
* Known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they have stable CNS disease for at least 4 weeks prior to the first dose of study drug and all neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids greater than 20 mg of prednisone daily for brain metastases (or the equivalent) for at least 7 days prior to trial treatment. All participants with carcinomatous meningitis are excluded regardless of clinical stability.
* Active cardiac disease as defined in protocol.
* Active chronic inflammatory bowel disease (ulcerative colitis, Crohn's disease) and participants with a history of bowel obstruction.
* Prior history of clinically significant bleeding, intestinal obstruction, or GI perforation within 6 months of enrollment.
* Must be at least 2 weeks beyond high dose systemic corticosteroids (however, low dose corticosteroids ≤10 mg prednisone or equivalent daily are permitted for reasons outside of CNS disease provided the dose is stable for 4 weeks).
* Active infection requiring systemic treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment. Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study
* Active autoimmune disease requiring systemic treatment with steroids or other immunosuppressive agent or any condition that in the Investigator's judgment precludes treatment with IPI-NIVO
* Received a live vaccine within 30 days prior to the first dose of study drug(s)
* History or evidence of interstitial lung disease (ILD) or non-infectious pneumonitis
* Known history of HIV-1/2 with uncontrolled viral load and on medications that may interfere with SN-38 metabolism.
* Known active Hepatitis B or Hepatitis C (In subjects with a history of HBV, hepatitis B core antibody (HBcAb) testing is required and if positive, then HB DNA testing will be performed and if positive the patient will be excluded).
* Other concurrent medical or psychiatric conditions that, in the Investigator's opinion, may be likely to confound study interpretation or prevent completion of study procedure and follow-up examinations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2021-04-30 (Actual); Primary Completion 2025-09-12 (Actual); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Maximum Tolerated Dose | Up to 12 months
  Determine the Maximum Tolerated Dose (MTD)/ Recommended Phase 2 dose (RP2D) of Sacituzumab Govitecan when combined with Ipilimumab and Nivolumab
Phase 2: Overall Response Rate | Up to 30 months
  Overall Response Rate (ORR) of Sacituzumab Govitecan with Ipilimumab and Nivolumab combination. ORR is defined as the rate of the best overall response as complete response (CR) or partial response (CR). OR will be summarized by the percentage of responses with a 95% confidence interval as calculated from Clopper-Pearson method.

SECONDARY OUTCOMES:
Phase 1: Overall Response Rate | Up to 12 months
  Overall Response Rate is defined as the rate of the best overall response as complete response (CR) or partial response (PR)
Phase 1: Duration of Response (DOR) | Up to 12 months
  Duration of Response will be calculated as the date of the first evaluation showing documented response, partial response (PR) or complete response (CR), to the date of the first progressive disease (PD) or death.
Phase 1: Progression Free Survival (PFS) | Up to 12 months
  Progression Free Survival defined as the time from start of treatment to the first event of death or progressive disease (PD) per RECIST 1.1.
Phase 2: Progression Free Survival (PFS) | Up to 30 months
  Progression Free Survival defined as the time from start of treatment to the first event of death or progressive disease (PD) per RECIST 1.1.
Phase 2: Duration of Response (DOR) | Up to 30 months
  Duration of Response will be calculated as the date of the first evaluation showing documented response, partial response (PR) or complete response (CR), to the date of the first progressive disease (PD) or death.
Phase 2: Overall Survival (OS) | Up to 30 months
  Overall Survival defined as the length of time from start of treatment until death by any cause. Participants will be evaluated using Kaplan- Meier estimation for survival for up to 6 months after discontinuation of study treatment; patients surviving longer than 6 months will be censored.

CONTACTS AND LOCATIONS:
Overall Officials: Jingsong K Zhang, MD, Principal Investigator — Moffitt Cancer Center; Guru Sonpavde, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/clinical-trials-research/clinical-trials/?source=footer